CLINICAL TRIAL: NCT06148922
Title: Brief Mental Health First Aid Program (bMHFA) for Parents to Improve Mental Health Literacy in Low-Income Families: A Three-Arm Cluster Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: bMHFA_low income family
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Issue
Keywords: Low-Income families; Parents; Mental Health First Aid (MHFA); brief intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Intervention group parents will receive a 2-hour workshop delivered by a registered nurse with a MHFA training certificate, in groups of up to 10 parents. Parents will receive a leaflet summarizing the training contents after the workshop. At 1 week and 1-, 3-, and 6-month follow-ups, the trained registered nurse will send a 5-minute reminder video via WhatsApp/WeChat to parents describing the key MHFA techniques. A set of online questionnaires will also be delivered to the parent-child dyads at these follow-ups.
  Interventions: Other: Brief Mental Health First Aid Workshop
- Control (No Intervention): The control group will receive no intervention. Only completing the sets of questionnaire.
- Intervention (Interview) (Other): Parents in the intervention group with the highest and lowest mental health literacy scores will be purposively invited to participate in one-to-one semi-structured interviews to explore their experience of the intervention.
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Brief Mental Health First Aid Workshop — a 2-hour workshop delivered by a registered nurse with a MHFA training certificate
  Arms: Intervention
Other: Semi-structured interviews — One-to-one, face-to-face semi-structured interviews will be conducted by a research assistant. The duration would be around 30 minutes.
  Arms: Intervention (Interview)

SUMMARY:
The goal of this Randomized Controlled Trial study is to test the effectiveness of the brief Mental Health First Aid Program (bMHFA) for parents to improve Mental Health Literacy in Low-Income families. The main questions it aims to answer are:

* Does the brief MHFA program improve mental health literacy among parents in low-income families?
* Does the brief MHFA program improve mental well-being among children in low-income families?

Participants will be randomly assigned to two groups, intervention and control group.

* Intervention group: attend a 2-hour training program on brief MHFA
* Intervention group: complete a set of questionnaire
* Intervention group: Interviews will be conducted at 12-month follow up
* Control: no need to attend any workshop
* Control: complete a set of questionnaire

DETAILED DESCRIPTION:
The traditional MHFA program covers many more mental disorders. Parents in the intervention group will receive a 2-hour workshop delivered by a registered nurse who has a MHFA training certificate from the Mental Health Association of Hong Kong. The first part includes an introduction that defines mental health and identifies mental health crises and symptoms, risk factors, and impacts. The second part of the workshop involves teaching parents the five key ALGEE techniques. The final part of the workshop concerns application of ALGEE in common types of mental disorders, including depression, anxiety, suicidal thoughts and behaviors, and substance abuse. Interviews will be held after 12-month of the intervention.

While the other group (control) will just have to complete a set of questionnaire, same set also need to complete by the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* able to speak Cantonese and read Chinese
* parenting at least one child aged 8-13 years
* receiving Comprehensive Social Security Assistance or have a household income less than the half of the median
* Children must be able to speak Cantonese and read Chinese

Exclusion Criteria:

* Parents and children with identified cognitive, behavioral, or mental problems will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 788 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Parents' level of mental health literacy | 12-month follow-up
  Chinese version of the mental health literacy scale

SECONDARY OUTCOMES:
Parents' level of mental health literacy | 1-week and 1-, 3-, and 6- month follow-ups
  Chinese version of the mental health literacy scale
Children's self-esteem | baseline and at the 1-week and 1-, 3-, 6-, and 12-month follow-ups
  Chinese version of the Rosenberg Self-Esteem Scale
Children's depressive symptoms | baseline and at the 1-week and 1-, 3-, 6-, and 12-month follow-ups
  Chinese version of the Center for Epidemiological Studies Depression Scale for Children
Children's anxiety symptoms | baseline and at the 1-week and 1-, 3-, 6-, and 12-month follow-ups
  Chinese version of the separation anxiety scale for children

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Katherine Lam, Phd, Principal Investigator — the polytechnic university of hong kong
Locations (1):
- The polytechnic university of Hong Kong, Hong Kong, Hong Kong